CLINICAL TRIAL: NCT00297154
Title: Lifestyle Modification in the Treatment of Heart Failure
Brief Title: The Effect of Diet and Exercise in Heart Failure
Acronym: LIMIT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Allison Pritchett, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-16557; K12RR017665 (NIH)
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure, Congestive; Metabolic Syndrome X; Obesity
Keywords: Heart failure, congestive; Metabolic Syndrome X; Obesity
MeSH Terms: conditions — Heart Failure; Metabolic Syndrome; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients continue receive a single educational session and continue medical managment of heart failure as per their physician
- Lifestyle modification (Experimental): Patients recieve weekly sessions with dietician, replace 2 meals/day with meal replacement beverage, and initiate a walking program.
  Interventions: Behavioral: Lifestyle Modification (diet, exercise, and behavior)

INTERVENTIONS:
Behavioral: Lifestyle Modification (diet, exercise, and behavior) — Patients recieve weekly sessions with dietician, replace 2 meals/day with meal replacement beverage, and initiate a walking program.
  Arms: Lifestyle modification

SUMMARY:
A growing number of people in this country are overweight or obese. This is concerning as increasing weight has been shown to increase the risk of developing heart failure. However, there is also research to suggest that in people who already have heart failure, heavier people live longer. So, how does being overweight put a person at risk for heart failure, but once they have heart failure, protect them? There is no clear explanation for this dilemma.

People who are obese commonly have other diseases, such as high blood pressure, high cholesterol, and diabetes, that increase the risk of developing heart disease. It is this group of diseases that is referred to as "The Metabolic Syndrome." People with the metabolic syndrome also have increased levels of inflammation and clotting proteins in their blood stream. Current treatment of the metabolic syndrome involves using medications for cholesterol, blood pressure, and diabetes. Diet and exercise are also commonly recommended.

"Lifestyle intervention programs" are programs that help people lose weight by changing their eating habits and exercise / activity routines. Weight loss and exercise have been shown to lower the risk of developing diabetes and improve diabetes control, improve cholesterol abnormalities, and lower blood pressure. These programs have not previously included heart failure patients, however.

We hypothesize that using a lifestyle intervention program in addition to the usual medications for heart failure will result in improved symptoms of heart failure and control of the metabolic syndrome.

This study will be the first research study to look at the use of diet and exercise in treating heart failure patients who are overweight / obese with "the metabolic syndrome." The study will last 6 months. From this study we hope to learn whether diet and exercise is helpful in treating heart failure patients who are overweight. Specifically, the study will look at the short term effects on cardiac risk factors (blood pressure, cholesterol, blood sugar), heart failure symptoms, and exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Must meet 3 or more of the NCEP defined criteria for metabolic syndrome

  * Waist circumference greater than 40 inches (102 cm) for men and 35 inches ( 88 cm) for women
  * Serum triglyceride level greater than or equal to 150 mg/dL
  * HDL level less than 40 mg/dL for men or 50 mg/dL for women
  * Blood pressure greater than 130/85 or treatment for hypertension
  * Fasting glucose greater than 110 mg/dL or treatment for diabetes
* Individuals with heart failure of ischemic or nonischemic etiologies * NYHA class II - III symptoms
* Left ventricular ejection fraction less than 40%
* Age 18-75 years
* BMI greater than 25 kg/m2
* Patients must have undergone a VO2 or exercise stress test within the last 6 months to exclude active ischemia or exercise-induced dysrhythmias

Exclusion Criteria:

* NYHA IV or 6 minute walk less than 300 meters
* Blood pressure greater than 160/100 mmHg
* Patients undergoing active titration of their cardiac medications
* Other comorbid illnesses which limit expected lifespan or affect the safety of interventions
* Weight loss of more than 10 pounds of non-edematous body weight within the past 3 months
* Pregnancy
* HIV+, active tuberculosis or hepatitis C
* Cancer requiring treatment within the past 5 years, unless the prognosis is excellent
* Unstable angina, myocardial infarction, coronary artery bypass surgery, or angioplasty within the last 3 months
* Angina with exertion
* History of malignant arrythmias (Ventricular Tachycardia / Ventricular Fibrillation) without implanted defibrillator
* Valvular heart disease:

  * Symptomatic aortic or mitral stenosis
  * Asymptomatic aortic or mitral stenosis that is moderate or greater in severity
  * Severe mitral regurgitation
* Hypertrophic cardiomyopathy
* Severe pulmonary hypertension with a pulmonary artery systolic pressure > 60 mmHg -
* Aortic aneurysm (>6 cm in diameter)
* Factors that may limit adherence to interventions or affect conduct of the trial

  * Unable or unwilling to given informed consent
  * Self-report of substance abuse within the past 12 months -
  * Failure to comply with the run-in dietary intake and exercise period
* History of bariatric surgery
* Chronic treatment with corticosteroids
* Current diagnosis of schizophrenia, other psychotic disorder, or bipolar disorder
* Current use of medications for weight loss
* Inability to walk two blocks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Measuring the change in Flow Mediated Dilation (FMD) and flow velocity integral (FVI) to assess endothelial function. | 6 months
Correlating change in vascular reactivity with renin, angiotensin II, and aldosterone levels. | 6 months

SECONDARY OUTCOMES:
Examining the impact of the lifestyle interventions on quality of life as measured by the validated Kansas City Cardiomyopathy Questionnaire. | 3 and 6 months
Assessing the effectiveness of the lifestyle intervention by sequential tracking of the weekly minutes of physical activity and body composition parameters. Overall exercise tolerance will be assessed using the 6 minute walk test. | 3 and 6 months
Defining alterations in metabolic syndrome parameters, inflammatory cytokines and platelet activation. | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allison M. Pritchett, M.D., Principal Investigator — Baylor College of Medicine; Douglas L Mann, M.D., Principal Investigator — Baylor College of Medicine